CLINICAL TRIAL: NCT02490332
Title: The Effects of Ventilation Tubes Versus no Ventilation Tubes for Recurrent Acute Otitis Media or Chronic Otitis Media With Effusion in 9 to 36 Month Old Greenlandic Children - a Randomised Clinical Trial
Brief Title: The Effects of Ventilation Tubes - The SIUTIT Trial
Acronym: SIUTIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to include the required number of participants
Sponsor: Zealand University Hospital (Other)
Collaborators: Government of Greenland, Agency for Health and Prevention (Unknown); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Malene Nøhr Demant, MD, PhD-student, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-112556
Record Dates: First submitted 2015-06-03; First posted 2015-07-03 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ventilation tube treatment (Experimental): Ventilation tube insertion in the tympanic membrane
  Interventions: Device: Ventilation tube treatment
- Conservative treatment (No Intervention): Conventional treatment

INTERVENTIONS:
Device: Ventilation tube treatment — Tympanostomy
  Other Names: Donaldson myringotomy tube
  Arms: Ventilation tube treatment

SUMMARY:
The prevalence of otitis media among Greenlandic children is one of the highest in the world and twenty per cent of schoolchildren have impaired hearing in the frequencies for normal speech. Yet, there are no national guidelines to ensure prevention and treatment of recurrent acute otitis media and chronic otitis media with effusion and impaired hearing in Greenlandic children. International studies from the developed part of the world have shown that otitis prone children may benefit from tubulation of the tympanic membrane. However, it is unknown if these results can be applied to Greenlandic children.

This PhD project will conduct a randomised controlled trial comparing tubulation of the tympanic membrane, in Greenlandic children aged 9-36 months with recurrent acute otitis media and/or chronic otitis media with effusion, to conservative treatment. The children will be followed for two years. Outcome measures will include number of visits to health clinics, number of tympanic membrane perforations, number of episodes with acute otitis media according to medical records, Quality of life, measured by the validated questionnaires OM6 and Caregiver Impact Questionnaire, number of episodes where per oral or intravenous antibiotics have been administered according to medical records and serious adverse events

The trial will be conducted in collaboration with the Greenlandic health authorities and Copenhagen Trial Unit.

With this trial the investigators hope to decrease the number of episodes with acute otitis media, the number of Greenlandic children with chronic perforations of the tympanic membrane and hearing impairment and increase quality of life.

The results will add important knowledge to the effect of ventilation tube treatment also in an international aspect. There are to date only less than a handful of high quality studies concerning this issue on an international basis. The study will be among the first addressing this problem among populations with high risk of otitis media and is also of interest to other indigenous populations and the developing part of the world.

ELIGIBILITY:
Inclusion criteria:

* Children aged 9-36 months.
* Children with at least one Greenlandic born parent with at least one Greenlandic born parent
* American Society of Anaesthesiologists physical status classification class 1 and 2
* B- or C2 - type curve measured by tympanometry at two visits three-four months apart or three episodes of acute otitis media in six months according to medical records or four episodes of acute otitis media in 12 months according to medical records
* Signed informed consent, signed by the legal guardian Exclusion criteria
* Children with orofacial cleft, Downs syndrome or known generalised immune deficiency
* American Society of Anaesthesiologists physical status classification class > 2.
* Lack of signed informed consent, signed by the legal guardian.

Description of experimental and control intervention Experimental intervention: The intervention group will be treated with bilateral Donaldson ventilation tubes administered in general anaesthesia Control intervention: The control intervention is based on the current practice in Greenland, which includes systemic antibiotic treatment as well as aural toilette and topical antibiotics. Ventilation tube insertion during the study period is not accepted in the control group.

Children in the intervention group as well as the control group will be seen once a year by the visiting ear-nose-and throat (ENT)-specialist and have a final consultation after at least two years after randomisation.

Ages: 9 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2016-02; Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
Number of visits to health clinic | Two years after randomisation
  Assessed by investigating medical records.

SECONDARY OUTCOMES:
Number of episodes of acute otitis media | Two years after randomisation
  According to medical records
Quality of life | Assessed at baseline, three months after randomisation, one year after randomisation, and at the end of the trial two years after randomisation
  Measured by validated questionnaires OM6 and Caregiver Impact Questionnaire
Number of episodes where per oral or intravenous antibiotics have been administered | Two years after randomisation
  According to medical records
Proportion of children with uni- or bilateral tympanic membrane perforations | Two years after randomisation
  Based on otoscopical photos, which will be anonymised and evaluated by an ENT-specialist without knowledge of the intervention

OTHER OUTCOMES:
Number of episodes of aural discharge | Two years after randomisation
  According to medical records
Serious adverse events | During the trial
  Any adverse event that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, or results in persistent or significant disability or incapacity.

CONTACTS AND LOCATIONS:
Overall Officials: Malene N Demant, MD, Principal Investigator — Køge University Hospital; Preben Homoe, MD, PhD, Study Director — Køge University Hospital
Locations (6):
- Greenland (6):
  - Aasiaat Regional Hospital, Aasiaat, Danmark
  - Ilulissat Regional Hospital, Ilulissat, Danmark
  - Nuuk Health Center, Nuuk, Danmark
  - Sisimiut Regional Hospital, Sisimiut, Danmark
  - Tasiilaq Health Center, Tasiilaq, Danmark
  - Qaqortoq Regional Hospital, Qaqortoq

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be publically available in depersonalised format after the end of trial on the Danish Data Archive and ZENODO.

REFERENCES:
- [Derived] MacKeith S, Mulvaney CA, Galbraith K, Webster KE, Connolly R, Paing A, Marom T, Daniel M, Venekamp RP, Rovers MM, Schilder AG. Ventilation tubes (grommets) for otitis media with effusion (OME) in children. Cochrane Database Syst Rev. 2023 Nov 15;11(11):CD015215. doi: 10.1002/14651858.CD015215.pub2. PMID 37965944
- [Derived] Demant MN, Jensen RG, Jakobsen JC, Gluud C, Homoe P. The effects of ventilation tubes versus no ventilation tubes for recurrent acute otitis media or chronic otitis media with effusion in 9 to 36 month old Greenlandic children, the SIUTIT trial: study protocol for a randomized controlled trial. Trials. 2017 Jan 19;18(1):30. doi: 10.1186/s13063-016-1770-x. PMID 28103950